CLINICAL TRIAL: NCT00995189
Title: A Clinical Evaluation of the Causes of Soft Contact Lens Related Dry Eye
Brief Title: Clinical Evaluation of the Causes of Contact Lens Related Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: M-09-03 / DRYS 1302 / IBIS
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2012-03

CONDITIONS: Contact Lens Related Dry Eye
Keywords: contact lens wear; multi-purpose solution; corneal staining
MeSH Terms: interventions — Contact Lenses

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OFR (Experimental): Opti-Free RepleniSH contact lens care solution used for 30 days
  Interventions: Device: Opti-Free RepleniSH; Device: Contact lenses
- RNM (Active Comparator): ReNu MultiPlus contact lens care solution used for 30 days
  Interventions: Device: ReNu MultiPlus; Device: Contact lenses

INTERVENTIONS:
Device: Opti-Free RepleniSH — Contact lens care solution containing polyquaternium-1 (PQT)
  Arms: OFR
Device: ReNu MultiPlus — Contact lens care solution containing polyhexamethylene biguanide (PHMB)
  Arms: RNM
Device: Contact lenses — Daily wear, frequent replacement contact lenses per participant's habitual brand and power.

SUMMARY:
The purpose of this study was to clinically evaluate the potential causes of contact lens-related dry eye.

DETAILED DESCRIPTION:
Daily wear soft contact lens wearers reporting significant contact lens-related dryness symptoms were enrolled. Late day dryness with contact lenses, intensity grade 3-5, frequency "sometimes / frequently / constantly" as evaluated by a questionnaire was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Reports late-day dryness symptoms with contact lens wear on questionnaire.
* Wears FDA Group 2 hydrogel, FDA Group 4 hydrogel, or silicone hydrogel lenses.
* Consistently uses either polyhexamethylene biguanide (PHMB) or polyquaternium-1 (PQT) contact lens care products (i.e. >6 months including 1 month immediately before enrollment).
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Wears daily disposable contact lenses.
* Has significant symptoms related to lens fit or lens deposits.
* Requires concurrent ocular medication (rewetting drops allowed).
* Has used Restasis® in the last 3 months.
* Wears punctal plugs fitted in the last 30 days.
* Has any current systemic or ocular abnormality, infection or disease.
* Uses any current systemic medication likely to affect tear film, e.g. antihistamines, betaadrenergic blockers, steroids.
* Has a history of refractive surgery.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Subjective Dryness | 2 weeks, one month

SECONDARY OUTCOMES:
corneal staining | 2 weeks, one month
conjunctival staining | two weeks, one month

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center For Trial Locations, Fort Worth, Texas, United States

REFERENCES:
- [Result] Chalmers RL, Young G, Kern J, Napier L, Hunt C. Soft Contact Lens-Related Symptoms in North America and the United Kingdom. Optom Vis Sci. 2016 Aug;93(8):836-47. doi: 10.1097/OPX.0000000000000927. PMID 27391535